CLINICAL TRIAL: NCT03258697
Title: The Pharmacokinetics and Effectiveness of Different Methods of Local LevoBupivacaine Injection, a Prospective Randomized Case Control Clinical Study on Primary Total Joint Replacement Model.
Brief Title: The Pharmacokinetics and Effectiveness of Local LevoBupivacaine Injection on Primary Total Joint Replacement Model.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201602050A3
Record Dates: First submitted 2017-08-16; First posted 2017-08-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2017-08

CONDITIONS: Arthropathy
Keywords: Local analgesia, Pharmacokinetics, Total joint replacement
MeSH Terms: conditions — Joint Diseases | interventions — Levobupivacaine

STUDY DESIGN:
Intervention Model Description: 1. PCA only
  2. Peri-articular Levobupivacaine + PCA
  3. Intra-articular Levobupivacaine + PCA
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patient blinded, observer blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patient-Controlled Analgesia (No Intervention): Patient had no local analgesic agent during total joint replacement. Patient had baseline Patient-Controlled Analgesia pump.
- Peri-articular LevoBupivacaine (Active Comparator): Patient had periarticular local analgesic agent, LevoBupivacaine Hydrochloride, during total joint replacement. Patient had baseline Patient-Controlled Analgesia pump.
  Interventions: Drug: Levobupivacaine Hydrochloride
- Intra-articular LevoBupivacaine (Experimental): Patient had intra-articular local analgesic agent, LevoBupivacaine Hydrochloride, during total joint replacement. Patient had baseline Patient-Controlled Analgesia pump.
  Interventions: Drug: Levobupivacaine Hydrochloride

INTERVENTIONS:
Drug: Levobupivacaine Hydrochloride — Different way of LevoBupivacaine injection
  Other Names: Chirocaine
  Arms: Intra-articular LevoBupivacaine; Peri-articular LevoBupivacaine

SUMMARY:
Total joint replacement is an ideal procedure to treat end stage joint disease. Good post-op pain relief could accelerate patient recovery and rehabilitation, and decrease admission days and medical cost. Local injection of LevoBupivacaine is an effective method in post-operative pain control. The effectiveness of local analgesia was noticed clinically. However, thorough studies about the pharmacokinetics of LevoBupivacaine, maintenance of effect, influence of post-operative rehabilitation are not well studied in different way of injection. The purpose of this study is to evaluate and analyze the pharmacokinetics and effect of local Levobupivacaine injection in different ways, the amount of post-operative fentanyl requirement after local injection, time to first fentanyl request, pain score, immediate post-operative function, side effect of analgesic agents, and medical cost, and to improve the quality of total joint replacement post-operative care.

DETAILED DESCRIPTION:
Single large dose of LevoBupivacaine had been proved good analgesic effect in total joint replacement surgery. However, the safety was not well studied. For better understanding the effect and safety of local analgesic agent, we choose LevoBupivacaine with different injection way to find out. We divide patient to three groups, for comparing the effectiveness of LevoBupivacaine, and safety of LevoBupivacaine by checking intra-blood concentration. The pre-emptive analgesics and post-operative analgesics were the same as routine protocol in other total joint replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Primary total joint replacement, no previous open surgery on the same joint
2. Age 50~80 y/o, Pre-operative diagnosis: degenerative osteoarthritis
3. Pre-operative deformity: varus <15°, valgus <15°, flexion contracture <15°.
4. Patients with normal heart function
5. Willing to receive post-operative questionnaire and outpatient clinic follow-up

Exclusion Criteria:

1. Allergy to Patient-Controlled Analgesia or LevoBupivacaine
2. Mental or cognitive illness that couldn't well response to questionnaire
3. American Society Anesthesiologist more than III degree
4. Liver cirrhosis, chronic renal insufficiency, heart disease or arrhythmia, insulin-dependent diabetes mellitus, and previous narcotic abuse history.
5. Not suitable for using patient-controlled analgesia pump by evaluation of anesthesiologist

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Dosage of analgesic opioid agent | post-operative day2
  The total dosage of opioid agent after local LevoBupivacaine injection

SECONDARY OUTCOMES:
Blood concentration of LevoBupivacaine | 25min, 90min, and coming morning after LevoBupivacaine injection
  Venous return of local LevoBupivacaine could cause the difference of blood concentration

OTHER OUTCOMES:
Functional score | Baseline, Post-operative day1, day2, week2, week6, week12, week24
  The difference of functional score

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chen Lo, M.S., Principal Investigator — Chang Gung Memorial Hospital, Linkou, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan, Taiwan

REFERENCES:
- [Background] Chen CC, Yang CC, Hu CC, Shih HN, Chang YH, Hsieh PH. Acupuncture for pain relief after total knee arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):31-6. doi: 10.1097/AAP.0000000000000138. PMID 25158837
- [Background] Chen DW, Hu CC, Chang YH, Lee MS, Chang CJ, Hsieh PH. Intra-articular bupivacaine reduces postoperative pain and meperidine use after total hip arthroplasty: a randomized, double-blind study. J Arthroplasty. 2014 Dec;29(12):2457-61. doi: 10.1016/j.arth.2013.12.021. Epub 2013 Dec 19. PMID 24439998
- [Background] Parvataneni HK, Shah VP, Howard H, Cole N, Ranawat AS, Ranawat CS. Controlling pain after total hip and knee arthroplasty using a multimodal protocol with local periarticular injections: a prospective randomized study. J Arthroplasty. 2007 Sep;22(6 Suppl 2):33-8. doi: 10.1016/j.arth.2007.03.034. Epub 2007 Jul 26. PMID 17823012
- [Background] Wasudev G, Smith BE, Limbird TJ. Blood levels of bupivacaine after arthroscopy of the knee joint. Arthroscopy. 1990;6(1):40-2. doi: 10.1016/0749-8063(90)90095-u. PMID 2310449
- [Background] Meinig RP, Holtgrewe JL, Wiedel JD, Christie DB, Kestin KJ. Plasma bupivacaine levels following single dose intraarticular instillation for arthroscopy. Am J Sports Med. 1988 May-Jun;16(3):295-300. doi: 10.1177/036354658801600317. PMID 3381989